CLINICAL TRIAL: NCT00554424
Title: A Randomised Controlled Trial of Intravaginal Lignocaine Injection Versus Placebo for Analgesia During Oocyte Recovery in an IVF Cycle
Brief Title: Local Anaesthetic for Transvaginal Egg Collection in IVF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Fertility Centre, New Zealand (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 01/12/180
Record Dates: First submitted 2007-11-03; First posted 2007-11-06 (Estimated); Last update posted 2007-11-06 (Estimated); Status verified 2007-11

CONDITIONS: Infertility
Keywords: oocyte retrieval; pain relief; Local anaesthetic
MeSH Terms: conditions — Infertility | interventions — Lidocaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LA (Active Comparator): Intravaginal and pre-peritoneal injection of 1% lignocaine into each side of the upper vagina under ultrasound guidance immediately prior to ultrasound guided transvaginal oocyte retrieval
  Interventions: Drug: lignocaine
- P (Placebo Comparator): Intravaginal saline placebo injection into each side of upper vagina under ultrasound guidance immediately prior to transvaginal oocyte retrieval
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: lignocaine — 20 mls of 1% lignocaine solution for injection, 10mls into each side of upper vagina, under ultrasound guidance immediately prior to transvaginal oocyte retrieval under ultrasound guidance from each ovary
  Arms: LA
Drug: normal saline — 20mls of normal saline solution, 10mls injected each side into upper vagina under ultrasound guidance, immediately prior to ultrasound guided transvaginal oocyte retrieval from each ovary
  Arms: P

SUMMARY:
The purpose of this study is to see whether injecting local anaesthetic into the vaginal tissues,just prior to transvaginal egg collection,will decrease the amount of pain experienced by women having their eggs collected on an IVF cycle. All women will also receive intravenous sedation as required as well as a sleeping tablet thirty minutes prior to the procedure which is our routine procedure for egg collection.

DETAILED DESCRIPTION:
Transvaginal oocyte retrieval is the most common method of oocyte collection in IVF cycles. A variety of different methods are used to provide analgesia/anesthesia for oocyte collection. Our unit has always used an oral pre-medication followed by intravenous fentanyl during the procedure but this doesn't seem to provide adequate analgesia for some women. The aim of this study was to compare the addition of intravaginal local anaesthetic injection versus saline placebo to our usual analgesia regime to see whether less intravenous fentanyl was required and whether the women experienced less pain during oocyte collection.

ELIGIBILITY:
Inclusion Criteria:

* About to undergo transvaginal oocyte retrieval

Exclusion Criteria:

* Already undergone oocyte retrieval and participated in study (i.e. 2nd or more oocyte collection procedure during study period)
* Allergy to lignocaine
* Oocytes only to be collected from one ovary
* Procedure expected to be exceptionally painful

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2002-03; Study Completion 2002-07 (Actual)

PRIMARY OUTCOMES:
Total dose of iv fentanyl used during oocyte collection | Length of oocyte collection (minutes)

SECONDARY OUTCOMES:
Pain score (cm on a Visual Analogue Scale) at 6 different points during oocyte collection | Actual point in time
Length of oocyte collection procedure | Time taken (minutes)
Occurence of nausea or vomiting | During oocyte collection procedure
Administration of atropine or anti -emetic | During oocyte collection procedure
Time spent in recovery room | Time from end of oocyte collection until discharge home
No of oocytes collected | During oocyte collection procedure
Number of oocytes fertilised | Assessed 18 hours after oocyte collection
Pregnancy outcome | 7 weeks gestation
Number of embryos frozen | Within 6 days of oocyte collection
Pulse rate at beginning and end of egg collection | Point in time
Maximum pulse rate during oocyte collection | Point in time during oocyte collection procedure

CONTACTS AND LOCATIONS:
Overall Officials: Sarah A Wakeman, FRANZCOG, Principal Investigator — The Fertility Centre
Locations (1):
- The Fertility Centre, Christchurch, Canterbury, New Zealand